CLINICAL TRIAL: NCT04587804
Title: Abdominal Treatment With Simultaneous Application of Noninvasive Repetitive Pulse Magnetic Stimulation (rPMS) and Radiofrequency
Brief Title: Abdomen - Fat Reduction and Muscle Toning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-703_100
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Fat Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Abdominal Toning and Reduction of Subcutaneous Fat (Experimental): simultaneous treatment by repetitive pulse magnetic stimulation and radiofrequency energy for toning of abdomen and reduction of subcutaneous fat
  Interventions: Device: rPMS+RF

INTERVENTIONS:
Device: rPMS+RF — The treatment administration phase will consist of three (3) treatments, delivered once a week. The applicator of the device will be applied over umbilicus and visible muscle contractions along with heating of the subcutaneous fat will be induced by the device.

SUMMARY:
This study will evaluate the clinical efficacy and safety of a simultaneous treatment by repetitive pulse magnetic stimulation and radiofrequency energy for toning of abdomen and reduction of subcutaneous fat. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete three (3) treatment visits and two to three follow-up visits. All of the study subjects will receive the treatment with the subject device.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of a simultaneous treatment by repetitive pulse magnetic stimulation and radiofrequency energy for toning of abdomen and reduction of subcutaneous fat. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete three (3) treatment visits and two to three follow-up visits. All of the study subjects will receive the treatment with the subject device.

At the baseline visit MRI will be performed, subject's weight and waist circumference will be recorded. Photos of the treated area will be taken.

The treatment administration phase will consist of three (3) treatments, delivered once a week. The applicator will be applied over umbilicus and visible muscle contractions along with heating of the subcutaneous fat will be induced by the device.

At the last therapy visit, the subject's weight and waist circumference will be recorded, and photos of the treated area will be taken. In addition, subjects will receive Subject Satisfaction Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE) including subject's experience of pain or discomfort after each procedure. Following each treatment administration and at all of the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

During the post-procedure visits (at 1-month and 3-month follow-up visits), the subjects will undergo MRI scanning. Also, subject's satisfaction will be noted and weight with waist circumference will be recorded. Photographs of the treated area will be taken. There will be an option of a 6-months follow-up visit, according to subject's availability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Voluntarily signed informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumour
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* Intrauterine device (IUD)
* Swollen or neoplastic tissues, space occupying lesions or skin eruptions in the treatment area
* Basedow's disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in adipose and muscular layer thickness between pre-treatment and post-treatment based on MRI scans | 4 months
  MRI will be conducted at the baseline visit and all follow-up visits. The imaging will be conducted at the same surface area each time.
  Hospital-grade MRI device will be used to scan abdominal area of each subject. The MRI scan without any contrast agent will be performed, with the scanned body segment determined by vertebrae T12 and S1. Lateral cuts from 5 cm below the umbilicus and 5 cm above the umbilicus will be evaluated for the thickness of muscle and subcutaneous adipose tissue.
Evaluation of change in adipose layer thickness between pre-treatment and post-treatment based on waist circumference measurements | 4 months
  Waist circumference measure will be conducted at the baseline visit, after last treatment and during follow-up visits.
  The waist circumference measure will be made at the top of the subject's iliac crest, with the tape held snugly, but not constricting, and at a level parallel to the floor. For the measurement, a stretch-resistant tape will be used.
  During the measuring, subject will stand with arms at the side, feet positioned close together, and weight evenly distributed across the feet. The subject will be instructed to relax and take a few deep, natural breaths before the actual measurement is made. The subjects will be measured in underwear only, after voiding the bladder.

SECONDARY OUTCOMES:
Evaluation of subject's satisfaction with the treatment using the Subject Satisfaction Questionnaire | 7 months
  The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome with answer "Strongly agree" being the most positive outcome and "Strongly disagree" the most negative. Subject satisfaction will be assessed after the last therapy visit and during the follow-up visits.
Safety of the device measured via the occurrence of adverse events or lack thereof | 7 months
  The occurrence of adverse events will be followed throughout the whole study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois